CLINICAL TRIAL: NCT06126380
Title: AT-1501-K209: BESTOW-EXTENSION: A Phase 2, Multicenter, Open-Label Extension Study to Evaluate the Long-Term Safety and Efficacy of Tegoprubart in Kidney Transplant Recipients
Brief Title: Long-Term Safety and Efficacy of Tegoprubart in Kidney Transplant Recipients
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Eledon Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AT-1501-K209; EU CTR (Other: 2023-503337-11-00); UTN (Other: U1111-1284-6127)
Record Dates: First submitted 2023-11-06; First posted 2023-11-13 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-03

CONDITIONS: Kidney Transplant Rejection
Keywords: Kidney Transplant; AT-1501; Renal Allograft Rejection; Prophylaxis; CD40L Inhibitor; Humanized blocking antibody to CD40L; monoclonal antibody; renal, transplant; ESRD; tegoprubart
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AT-1501 (Experimental): AT-1501 20 mg/kg administered every 3 weeks IV + MMF 1000 mg per os (orally) (PO) twice daily (BID) or MPS 720 mg PO BID + Corticosteroids 5 mg of prednisone PO once daily (QD) or equivalent
  Interventions: Drug: AT-1501
- Tacrolimus (Active Comparator): Tacrolimus dosed PO BID with the dose titrated to maintain a trough concentration of 6-8 ng/mL+ MMF 1000 mg PO BID or MPS 720 mg PO BID + Corticosteroids 5 mg of prednisone PO QD or equivalent
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: AT-1501 — AT-1501 20 mg/kg administered every 3 weeks IV + MMF 1000 mg PO twice daily (BID) or MPS 720 mg PO BID + Corticosteroids 5 mg of prednisone PO once daily (QD) or equivalent
  Other Names: Tegoprubart
  Arms: AT-1501
Drug: Tacrolimus — Tacrolimus dosed PO BID with the dose titrated to maintain a trough concentration of 6-8 ng/mL+ MMF 1000 mg PO BID or MPS 720 mg PO BID + Corticosteroids 5 mg of prednisone PO QD or equivalent
  Arms: Tacrolimus

SUMMARY:
This study will evaluate the long term safety and efficacy of AT-1501 (tegoprubart) compared with tacrolimus in patients undergoing kidney transplantation.

DETAILED DESCRIPTION:
This is a multicenter, open-label, active control extension study to assess the long-term safety and efficacy of AT-1501 (tegoprubart) compared with tacrolimus in the preservation of allograft function after kidney transplantation.

The number of patients enrolled for OLE study will depend on the enrollment in the Parent studies. To be eligible for participation in this study, participants must have completed a designated Parent study.

Participants in this study will continue the treatment regimen they were receiving in the Parent study. Dose regimens will include either AT-1501 (tegoprubart) or tacrolimus.

ELIGIBILITY:
Inclusion Criteria:

* Successfully completed qualifying Parent study, where entry into the OLE was offered;
* Continue to be able to understand the key components of the study as described in the written ICF, and is willing and able to provide written informed consent;
* Agree not to participate in another interventional study while on treatment;
* If female, is surgically sterile or 2 years postmenopausal. Women of childbearing potential may be enrolled if a pregnancy test is negative at baseline. Women of childbearing potential and men with partners that are of childbearing potential must agree to use highly effective methods of contraception from baseline, through 90 days after the last administration of the study drug. Examples of acceptable methods of contraception are described in Table 6.
* If male, agree to use a medically accepted highly effective method of contraception and agree to use this method for 90 days after last administration of the study drug and agree to not donate sperm for 90 days after last administration of the study drug.

Exclusion Criteria:

* Unwilling or unlikely to comply with the study requirements, in the opinion of the Investigator;
* Met any of the stopping criteria or discontinued study drug in the Parent study;
* Pregnant or breastfeeding.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability - Incidence of Treatment Emergent Adverse Events | Assessed from date of enrollment through Month 48
  Incidence of treatment-emergent serious adverse events (TESAEs), treatment-emergent adverse events (TEAEs), and treatment-emergent AEs of special interest (TEAEoSI).
Safety and Tolerability - Kidney Transplant Medication Side Effects | Assessed from date of enrollment through Month 48
  Kidney transplant medication side effects using the Modified Transplant Symptom Occurrence and Symptom Distress Scale-59 (MTSOSD) at baseline and 12, 24, 36, and 48 months.

SECONDARY OUTCOMES:
The proportion of patient and graft survival at 12, 24, 36, and 48 months | Assessed from date of enrollment through Month 48
  A participant is considered to have graft functional impairment if they have an eGFR <60 mL/min/1.73m^2.
The proportion of participants with Graft function impairment at 12, 24, 36, and 48 months | Assessed from date of enrollment through Month 48
  A participant is considered to have graft functional impairment if they have an eGFR <60 mL/min/1.73m^2.
Proportion of participants with BPAR at 12, 24, 36, and 48 months | Assessed from date of enrollment through Month 48
  The Proportion of participants with BPAR at 12, 24, 36, and 48 months.
Proportion of composite endpoint (graft failure, BPAR, or death) at 12, 24, 36, and 48 months | Assessed from date of enrollment through Month 48
  The Proportion of participants with composite endpoint (graft failure, BPAR, or death) at 12, 24, 36, and 48 months.

CONTACTS AND LOCATIONS:
Locations (43):
- United States (26):
  - University of California Los Angeles, Los Angeles, California
  - Keck School of Medicine of USC, Los Angeles, California
  - University of California, Irvine Medical Center, Orange, California
  - University of California, Davis Medical Center, Sacramento, California
  - Jacobs Medical Center at UC San Diego Health, San Diego, California
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Tampa General Hospital, Tampa, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - University of Chicago, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Tulane Medical Center, New Orleans, Louisiana
  - John Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University in St. Louis, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - New York University Langone Health - Tisch Hospital, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - University of Pittsburgh Medical Center, Harrisburg, Pennsylvania
  - UT Southwestern, Dallas, Texas
  - Virginia Commonwealth University, Richmond, Virginia
- Australia (2):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Fiona Stanley Hospital, Perth, Western Australia
- Brazil (2):
  - Fundação Oswaldo Ramos - Hospital do Rim, São Paulo
  - Hospital das Clínicas da Faculdade de Medicina de São Paulo, São Paulo
- Canada (2):
  - St. Paul's Hospital, Vancouver, British Columbia
  - McGill University Health Care Centre, Montreal, Quebec
- France (4):
  - Groupe Hospitalier Pellegrin, Bordeaux
  - CHU Grenoble-Alpes - Hopital Nord Michallon, Grenoble
  - Centre Hospitalier Universitaire Dupuytren, Limoges
  - CHU de Toulouse - Hopital de Rangueil, Toulouse
- Charite Universitatsmedizin Berlin, Berlin, Germany
- Spain (5):
  - Hospital del Mar - Parc de Salut Mar, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinical de Barcelona, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Germans Trias i Pujol, Barcelona
- Oxford University Hospitals NHS Foundation Trust - John Radcliffe Hospital, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No